CLINICAL TRIAL: NCT02928276
Title: Prediction of the Response to Anti-TNFs DMARDs Based on the RheumaKit ® Platform (RK-Tx-01)
Brief Title: Predictive Analytics for Theranosis in RA
Acronym: PAnTheRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DNAlytics (Industry)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RK-Tx-01
Record Dates: First submitted 2016-09-06; First posted 2016-10-10 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumakit; Rheumatoid Arthritis; anti-TNF
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All eligible patients
  Interventions: Other: RheumaKit: Prediction of the response to anti-TNFs DMARDs

INTERVENTIONS:
Other: RheumaKit: Prediction of the response to anti-TNFs DMARDs

SUMMARY:
RA is the most common inflammatory, persistent and progressive disease of the joints with serious co-morbidities and huge health and socio-economic impact worldwide.

DETAILED DESCRIPTION:
The current standard therapeutic strategy for RA patients is to initiate a DMARDs therapy, (e.g. MTX) with serious side effects. This also applies to some PSO or SNSA patients. MTX is however inefficient in about 40% of the cases. Other treatments (biological DMARDs) must thus be initiated, which have an overall similar effectiveness and side effects and an higher cost (around 13kEUR/year/patient). Therapeutic choices are based on symptoms and blood tests including markers of inflammation which are inadequate to predict disease evolution and response to treatments. Improving RA management requires to improve the adequacy of the therapeutic strategies. The earlier the disease is correctly addressed, the more likely its progression and irreversible damages to the joints will be limited. DNAlytics recently developed RheumaKit a differential diagnostic solution for UA patients. UA is a condition in which joint inflammation is present, but a precise diagnosis cannot be made, due to the lack of sensitivity of presently available diagnostic techniques. RheumaKit is a multi-gene expression solution that discriminates RA from other joint conditions. A diagnostic model train to identify patients suffering from RA, SNSA or OA. RheumaKit diagnostic accuracy is higher than 90%, a performance that is better than any other diagnostic solution designed until now, including the ACR/EULAR 2010 criteria for the diagnosis of RA. See working principle below. Beyond diagnosis, DNAlytics wants to make RheumaKit evolve towards treatment recommendation applications (theranostic applications) for patients eligible for biological DMARDs. On one hand, the diseases of these patients have been more and more described in terms of the activity of several metabolic pathways (T & B cells activation, Extra cellular matrix, Inteferon, TNF). On the other hand, the existing treatments also have been more and more described in terms of the pathways they target. The RheumaKit signature contains many markers that are representative of these pathways of interest. RheumaKit thus now provides a snapshot of the activity of seven metabolic pathways known from literature to be related to diseases mechanisms, or to be target of existing treatments. In this study, DNAlytics wants to show that based on a score defined on the RheumaKit platform, the response or non- response to anti-TNFs, representing the largest category of biological DMARDs, can be predicted before treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all of the following criteria:

* Signed the ICF and covered by health insurance.
* At least 18 years old.
* For women, use of a reliable method of birth control or remain abstinent during the study, or have had surgical sterilization or women above 60 years of age.
* Having undergone at least 3 months of synthetic DMARD treatment while being strictly eligible for it (diagnosed with RA) and being at a stable dose at least for the last month, and showing no satisfactory response to this therapy.
* Be eligible for biological DMARD treatment according to local regulation and practice.
* Willing and able to comply with scheduled visits, treatment plan, tests and other protocol procedures.

Exclusion Criteria:

Patients must satisfy none of the following criteria:

* Arthritis history longer than 5 years.
* Biological DMARD therapy already initiated.
* Be diagnosed with septic arthritis.
* Be pregnant or breastfeeding/lactating women.
* Diagnosed with HIV, hepatitis B, hepatitis C, Crohn's disease, fibromyalgia.
* Diagnosed with other inflammatory arthritic syndrome than RA.
* have a chronic pain condition that would confound evaluation of the patient.
* Be identified as at too high risk for biopsy or for biologic therapy.
* Be identified as having psychological, familial, social or geographical conditions which could potentially hamper compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-12 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Ability of a score | Up to 12 months
  To show the ability of a score, computed prior to treatment initiation, to be predictive of the individual anti-TNF response. The score is based on the RheumaKit transcriptomic profiles from a set of small synovial biopsies from a given joint also harvested before anti-TNF treatment initiation.

SECONDARY OUTCOMES:
Identify additional/alternative mappings | Up to 12 months
  To identify additional/alternative mappings between components of gene expression profiles obtained via the RheumaKit assay (extended, and possibly combined to clinical and biological information) and efficacy of anti-TNFs biological DMARDs.
Validate the sample logistics at an international scale. | Up to 12 months
  To validate the feasibility of the implementation of a molecular biology test in rheumatology based on synovial tissue at an international scale. This covers both logistics and patient agreeableness aspects.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Durez, MD, PhD, Principal Investigator — Clinique Universitaire Saint-Luc
Locations (5):
- Belgium (4):
  - Clinique Universitaires Saint-Luc, Brussels, Bruxelles-capital
  - CHU Saint-Pierre, Brussels
  - UZLeuven, Gasthuisberg, Leuven
  - CHU Liège, Liège
- Parc Taulí Hospital Universitari, Sabadell, Catalunia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lauwerys BR, Hernandez-Lobato D, Gramme P, Ducreux J, Dessy A, Focant I, Ambroise J, Bearzatto B, Nzeusseu Toukap A, Van den Eynde BJ, Elewaut D, Gala JL, Durez P, Houssiau FA, Helleputte T, Dupont P. Heterogeneity of synovial molecular patterns in patients with arthritis. PLoS One. 2015 Apr 30;10(4):e0122104. doi: 10.1371/journal.pone.0122104. eCollection 2015. PMID 25927832